CLINICAL TRIAL: NCT00398619
Title: A Double-blind, Placebo Controlled Pharmacodynamic Study of the Effect of INCB013739 on Systemic and Adipose Tissue 11βHSD1 Activity in Obese, Insulin Resistant Subjects.
Brief Title: A Study of the Effect of INCB013739 on Cortisone Reducing Enzyme Activity in Obese People Predisposed to Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: William Williams, M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB13739-103
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — INCB 13739

INTERVENTIONS:
Drug: INCB13739

SUMMARY:
The purpose of this study is to determine whether the investigational drug INCB013739 has an effect on systemic and adipose tissue 11-HSD1 activity in obese, insulin resistant subjects.

DETAILED DESCRIPTION:
"Proprietary Information: Exploratory (Non-Confirmatory) Trial".

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 years and 65 years of age.
* BMI between 30 and 42 kg/m2, inclusive.
* FPG <126 mg/dL

Exclusion Criteria:

* Meet criteria for diagnosis of diabetes mellitus at the screening evaluation, female subjects with a history of gestational diabetes are permitted.
* Are receiving oral antidiabetic agents within the 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacokinetics of INCB013739 through analysis of blood samples. | Serial collections at each visit
Evaluation of change in cortisol laboratory values | Serial collections at each visit
Assessment of ECGs, laboratory results and physical exams for adverse events | Measured from baseline through study completion

CONTACTS AND LOCATIONS:
Overall Officials: William V Williams, MD, Study Director — Incyte Corporation
Locations (2):
- United States (2):
  - Beverly Hills, California
  - Chula Vista, California